CLINICAL TRIAL: NCT03143400
Title: Behavior of Various Galenic Forms of a Probiotic in the Digestive Tract
Acronym: PROBIOSIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: 3i nature (Other); European Regional Development Fund (Other); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHU-322; 2016-A00597-44 (Other: 2016-A00597-44)
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Healthy Volunteer; Terminal Ileostomy
Keywords: Probiotics; Galenic form; Digestive tract; Intestinal microbiota; Lactobacillus salivarius

STUDY DESIGN:
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy volunteers (Active Comparator): Healthy volunteers will test each of the 3 galenic forms of Lactobacillus salivarius on 3 periods of 7 days. Each period will be separated from another with a 14-day wash-out period at least.
  Interventions: Drug: Lactobacillus salivarius BL 3123
- Ileostomized patients (Active Comparator): Ileostomized patients will only take a unique dose of each probiotic. Each intake of a different probiotic will be separated from another by a 14-day wash-out period at least.
  Interventions: Drug: Lactobacillus salivarius BL 3123

INTERVENTIONS:
Drug: Lactobacillus salivarius BL 3123 — Two classic forms will be tested (powder and pill). An innovative galenic form (pill with retarded release), developed to enhance intestinal viability and probiotic efficacy, will also be tested.

SUMMARY:
The aim of this study is to assess the behavior of a model probiotic strain, Lactobacillus salivarius, in the digestive tract of healthy volunteers and of ileostomized patients, depending on its galenic form.

Two classic forms will be tested (powder and pill). An innovative galenic form (pill with retarded release), developed to enhance intestinal viability and probiotic efficacy, will also be tested.

DETAILED DESCRIPTION:
Probiotic survival in the stomach and in stools will be assessed on 9 healthy volunteers. It will be evaluated in the stomach after one unique probiotic intake. Gastric content will be collected at different times, up until an hour after probiotic ingestion.

Fecal probiotic survival will be evaluated after a 7-day period of probiotic intake. Initial stool collection, before first probiotic intake, will be used as control. Stools will be collected after 7 days of treatment (D8) and 3 days after last intake (D10).

Probiotic survival in the small intestine will be assessed on 9 patients with stable medical condition that either have a terminal or preterminal ileostomy. It will be evaluated after one unique probiotic intake. Ileal content will then be collected within 4 hours after intake.

Probiotic survival will be evaluated in the stomach, small intestine and in stools by qPCR and determination of CFU. Microbiota composition will be determined by pyrosequencing on ileal and fecal samplings. Finally, metabolic activity will be determined by chromatography with a short chain fatty acid dosage.

Healthy volunteers will test each of the 3 galenic forms of Lactobacillus salivarius on 3 periods of 7 days. Each period will be separated from another with a 14-day wash-out period at least.

Ileostomized patients will only take a unique dose of each probiotic. Each intake of a different probiotic will be separated from another by a 14-day wash-out period at least.

ELIGIBILITY:
Inclusion Criteria:

For the healthy volunteer group :

* age between 18 and 65 years old
* without previous digestive pathology that could have modified probiotic survival either by the disease itself or by its treatments (IBD, cholestatic disease, pancreatic insufficiency)
* without previous digestive surgery (except from appendectomy)
* ability to sign written informed consent
* health insurance

For the patients with a ostomy pouch :

* Age between 18 and 65 years old
* Terminal or preterminal (less than 30 cm of resected ileon) ileostomy performed more than 2 months ago with a stabilized digestive situation and a healthy residual intestine.
* Without other digestive resection (gall bladder, stomach, pancreas)
* Healthy and diversified diet
* Health insurance

Exclusion Criteria for both groups :

* Acute disease, digestive in particular
* Intake of antibiotics and non-steroidal anti-inflammatory drugs in the last 3 months
* Intake of probiotics and symbiotic within the month before inclusion, either in a food supplement form (Lactibiane, Probiolog, Bacilor, Ergyphyllus, Bion3,) or as a milk product (Actimel, Activia, LC1)
* Intake of an antacid or gastric antisecretory (anti-H2, proton pump inhibitor) the week before study
* Intake of gastric emptying modificators and drugs that could slow down bowel movement (domperidone, metoclopramide, morphinise, loperamide) within 48 hours before study.
* Pregnant or breastfeeding women
* Patient under guardianship or curatorship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Survival rate of Lactobacillus salivarius | 7 days
  Measured by qPCR and determination of CFU in gastric content and in stools for each galenic form.

SECONDARY OUTCOMES:
Probiotic residual amount in control healthy volunteer | 10 days
  Measured by qPCR and determination of CFU
Probiotic residual amount in ostomy pouch | 8 days
  Measured by qPCR and determination of CFU. Fecal microbiota composition at D0 and D8 after the first intake, in the healthy volunteer group, for each 3 galenic forms.
Ileal microbiota composition | 8 days
  Patients with ostomy pouch
Potential occurrence of digestive symptoms or extra-digestive | 8 days
  Nausea, bloating, flatulence, abdominal pain, intestinal transit modification
Comparison of residual probiotic amount between in vivo and in vitro collection in the stomach, ileon and in stools | 8 days
  Measured by qPRC and determination of CFU number

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France